CLINICAL TRIAL: NCT00604188
Title: A Randomized Acceptability and Safety Study of Suboxone Induction in Heroin Users
Brief Title: A Randomized Acceptability and Safety Study of Suboxone Induction in Heroin Users (P05042)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05042
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Opiate Dependence; Drug Dependence; Substance Dependence
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Direct Suboxone Induction (Experimental): Participants received 8 mg of Suboxone and placebo Subutex on Day 1, 16 mg of Suboxone and placebo Subutex on Day 2, and all participants received open label Suboxone from Day 3 to Day 28. Suboxone dosage may be titrated from Day 4 to Day 28 up to 24 mg per day.
  Interventions: Drug: Suboxone (SCH 000484)
- Subutex-to-Suboxone Induction (Active Comparator): Participants received 8 mg Subutex and placebo Suboxone on Day 1, 16 mg Subutex and placebo Suboxone on Day 2, and all participants received open label Suboxone from Day 3 to Day 28. Suboxone dosage may be titrated from Day 4 to Day 28 up to 24 mg per day.
  Interventions: Drug: Suboxone (SCH 000484); Drug: Subutex (SCH 028444)

INTERVENTIONS:
Drug: Suboxone (SCH 000484) — 2 mg and 8 mg sublingual tablets, Contains Buprenorphine Hydrochloride and Naloxone. Daily dosage of 8 mg - 24 mg. Duration: 28 Days
  Other Names: SCH 000484
Drug: Subutex (SCH 028444) — 2 mg and 8 mg sublingual tablets, Contains Buprenorphine Hydrochloride. Daily dosage of 8 mg - 24 mg. Duration: 28 Days
  Other Names: SCH 028444
  Arms: Subutex-to-Suboxone Induction

SUMMARY:
The purpose of this study is to assess the acceptability and safety of Suboxone in heroin users as a replacement therapy for opioid dependency by comparing the clinical response of participants who are inducted directly onto Suboxone with that of participants who are inducted first to Subutex and then transferred to Suboxone.

DETAILED DESCRIPTION:
Rationale: Once Suboxone becomes available for widespread clinical use, it is anticipated that opioid-dependent patients seeking treatment with buprenorphine will be placed directly onto Suboxone. Two strategies that have had good success for inducting patients onto Suboxone have been developed: 1) a "bridging" procedure in which patients initiate therapy with Subutex and then transfer to Suboxone, and 2) a direct Suboxone induction procedure. However, there have been no controlled studies of direct Suboxone induction, and it is not clear whether using a Subutex-to-Suboxone induction procedure would produce any added clinical benefit for the patient relative to direct Suboxone induction.

This study addresses a post-marketing commitment to the European Medicines Agency to conduct a prospective, controlled study of induction with Suboxone. Using a prospective, randomized, active-drug-controlled, double-blind and double-dummy design, this study will assess the acceptability and safety of Suboxone in heroin users by comparing the clinical response of participants who are inducted directly onto Suboxone with that of participants who are inducted first to Subutex and then transferred to Suboxone. The dose regimen used during the induction phase of this study is identical to that used in the pivotal efficacy study comparing Suboxone and Subutex (Fudala et al, 2003), which is included in the Suboxone Summary of Product Characteristics. The data collected in this study will include information on the extent of opioid use before treatment initiation.

Two strategies for inducting opioid-dependent patients using short-acting opioids (eg, heroin) onto Suboxone have emerged from published US studies. One involves using Subutex to "bridge" the transition to Suboxone by using Subutex over the first 2 days before transferring directly to Suboxone on the third day. The other involves direct Suboxone induction, in which patients receive Suboxone as the initial dose followed by continued rapid Suboxone dose titration.

In the pivotal efficacy study, opiate-dependent heroin users assigned to either Subutex or Suboxone groups received an induction dose of 8 mg of Subutex (administered as a single 8-mg tablet) on Day 1 and 16 mg of Subutex (administered as two 8-mg tablets) on Day 2. The 109 participants assigned to Suboxone received 16 mg of Suboxone (administered as two 8-mg tablets) on Day 3, and the 105 participants assigned to Subutex received 16 mg of Subutex (administered as two 8-mg tablets) on Day 3. The induction schedule used in the pivotal trial, in which a Subutex-to-Suboxone bridging procedure was used, was successful for inducting heroin-dependent patients onto Suboxone, achieving good compliance and resulting in relatively few AEs accounting for treatment discontinuation.

Overall, several large-scale studies using Suboxone as an initial medication have been conducted with good results, and it appears clear that, as was the case in the pivotal study, most patients safely tolerate a total dose of at least 8 mg on the first day of treatment. However, as these studies were not controlled, it remains unclear whether using a Subutex-to-Suboxone induction procedure would produce any added clinical benefit to the patient relative to a direct Suboxone induction procedure. Furthermore, there have been no studies of direct Suboxone induction outside of the United States.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be males or non-pregnant, non-lactating females.
* Participants must be at least 15 years of age, of either sex, and any race.
* Participants (and/or the parent or guardian for participants under the age of legal consent or who otherwise are unable to provide independent consent) must demonstrate willingness to participate in the study and to adhere to dose and visit schedules.
* Participants must meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for opioid dependence.
* Participants must have a methadone- and buprenorphine-negative UDS result prior to randomization.
* Each participant must confirm that he or she is practicing adequate contraception. Female volunteers of childbearing potential (including women who are less than 1 year postmenopausal and women who will be sexually active during the study) must agree to use a medically accepted method of contraception or must be surgically sterilized prior to screening, while receiving protocol-specified medication, and for 30 days after stopping the medication. Women who have been postmenopausal for >=1 year (ie, women who have experienced 12 or more consecutive months of amenorrhea) will be exempted from the requirement to use contraception during the study. Acceptable methods of contraception include condoms (male and female) with or without a spermicidal agent, diaphragm or cervical cap with a spermicidal agent, medically prescribed intrauterine device, oral or injectable hormonal contraceptives, and surgical sterilization (eg, hysterectomy or tubal ligation).
* Female participants of childbearing potential must have a negative urine beta-human chorionic gonadotropin (beta-hCG) test prior to enrollment in the study

Exclusion Criteria:

* Participants for whom treatment with either Subutex or Suboxone as required in the protocol would be inconsistent with national labeling.
* Participants who are unwilling or unable to comply with the requirements of the protocol (eg, pending incarceration) or are in a situation or condition that, in the opinion of the investigator, may interfere with participation in the study.
* Participants who are participating in any other clinical study in which medication(s) are being delivered.
* Participants with known allergy or sensitivity to buprenorphine or naloxone.
* Participants who are on the staff, affiliated with, or a family member of the staff personnel directly involved with this study.
* Participants with serious untreated Axis I DSM-IV-TR psychiatric co-morbidity (eg, those who are actively suicidal or homicidal, have untreated schizophrenia, etc). Polysubstance abuse or dependence will not exclude participants except in the case of unauthorized and significant benzodiazepine use requiring medical detoxification or alcohol dependence requiring medical detoxification.
* HIV-positive participants with clinical acquired immunodeficiency syndrome (AIDS).
* Methadone or buprenorphine maintenance or detoxification within 30 days of enrollment.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2008-02-22 (Actual); Primary Completion 2009-12-10 (Actual); Study Completion 2009-12-10 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Amass L, Pukeleviciene V, Subata E, Almeida AR, Pieri MC, D'Egidio P, Stankova Z, Costa A, Smyth BP, Sakoman S, Wei Y, Strang J. A prospective, randomized, multicenter acceptability and safety study of direct buprenorphine/naloxone induction in heroin-dependent individuals. Addiction. 2012 Jan;107(1):142-51. doi: 10.1111/j.1360-0443.2011.03577.x. Epub 2011 Oct 12. PMID 21749526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 188 participants were recruited in this study.
Pre-assignment Details: 188 participants were randomized in the study; however one did not receive any study medication. Therefore the intent-to-treat (ITT) population was 187 participants.
Period: Overall Study
Arm/Group | Direct Suboxone Induction | Subutex-to-Suboxone Induction
Started | 93 | 95 (The ITT population for Subutex-to-Suboxone Induction is 94 participants)
Completed | 66 | 70
Not Completed | 27 | 25
Not completed — Adverse Event | 1 | 4
Not completed — Lost to Follow-up | 17 | 15
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Non-compliance with protocol | 4 | 4
Not completed — Did not receive study drug | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Direct Suboxone Induction | Subutex-to-Suboxone Induction | Total
Number analyzed (Participants) | 93 | 94 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (8.4) | 30.5 (8.2) | 30.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 46
  Male | 72 | 69 | 141

OUTCOME MEASURES:

1. Primary Outcome: Responders at Day 3
Description: Responders included the number of participants who received the scheduled dose of Suboxone at the Day 3 study visit. Participants who discontinued the study at Day 3 were considered non-responders.
  All participants that continued the study received Suboxone tablets on Day 3.
Time Frame: 3 days
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | Direct Suboxone Induction | Subutex-to-Suboxone Induction
Number analyzed (Participants) | 93 | 94
Participants
  Responders | 85 | 85
  Non responders | 8 | 9

2. Secondary Outcome: Illicit Opioid and Non-opioid Drug Use: Urine Drug Screen (UDS)
Description: Number of participants who tested negative on UDS during open-label phase on Day 28. The drugs screened on Day 28 included amphetamines, methamphetamines, cocaine, morphine, methadone, benzodiazepines, and tetrahydrocannabinol. Buprenorphine was only tested at screening and randomization according to protocol, therefore no values for buprenorphine are available for Day 28.
Time Frame: 28 days
Population: Participants with missing data were not included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Direct Suboxone Induction | Subutex-to-Suboxone Induction
Number analyzed (Participants) | 79 | 82
Participants
  Tetrahydrocannabinol | 65 | 59
  Cocaine | 70 | 69
  Amphetamines | 77 | 81
  Benzodiazepines | 59 | 64
  Methamphetamines | 79 | 80
  Morphine | 66 | 67
  Methadone | 76 | 81
  Buprenorphine | NA — Per protocol, buprenorphine testing was not performed on Day 28. | NA — Per protocol, buprenorphine testing was not performed on Day 28.

3. Secondary Outcome: Illicit Opioid and Non-opioid Drug Use: Substance Use Inventory (SUI)
Description: Number of participants with intravenous use of drug as measured by self-reported SUI from Days 3-28. The SUI form consisted of questions addressing the number of days and times a drug was used, and the route of drug use. For suboxone the use of scheduled study medication was not considered illicit use.
Time Frame: Days 3 to 28
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | Direct Suboxone Induction | Subutex-to-Suboxone Induction
Number analyzed (Participants) | 93 | 94
Participants
  Subutex - Non prescription source | 0 | 0
  Suboxone - Non prescription source | 0 | 0
  Suboxone - Illicit use from study supplies | 0 | 0
  Heroin | 12 | 14
  Other opioids | 0 | 0
  Methadone | 0 | 0
  Methamphetamine | 0 | 0
  Cocaine | 2 | 4
  Benzodiazepines/Tranquilizers | 0 | 0

4. Secondary Outcome: Self-reported Opioid Withdrawal Symptoms (SOWS)
Description: SOWS were 16 items whose intensity was scored on a scale from 0 (not at all) to 4 (extremely) for a maximum possible score of 64. A total score of 0 represented the best outcome and a score of 64 represented the worst outcome. Participants were scored for SOWS at baseline (prior to randomization) and on Day 28. Reported are the scores for Day 28, and the change in scores from baseline to Day 28.
Time Frame: Baseline and 28 days
Population: Participants with SOWS data reviewed for completeness and within visit date consistency were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Direct Suboxone Induction | Subutex-to-Suboxone Induction
Number analyzed (Participants) | 69 | 72
Score on a scale
  Score on Day 28 | 3.8 (6.77) | 3.4 (5.95)
  Change from Baseline to Day 28 | -23.3 (14.1) | -21.9 (13.4)

5. Secondary Outcome: Observer-rated Opioid Withdrawal Symptoms (OOWS)
Description: The OOWS were 13 physically observable signs that were present (scored 1) or absent (scored 0). A total score of 0 represented the best outcome and a total score of 13 represented the worst outcome. Participants were scored for OOWS at baseline (prior to randomization) and on Day 28. Reported are the total score for Day 28, and the change in scores from baseline to Day 28.
Time Frame: Baseline and 28 days
Population: Participants with OOWS data reviewed for completeness and within visit date consistency were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Direct Suboxone Induction | Subutex-to-Suboxone Induction
Number analyzed (Participants) | 69 | 72
Score on a scale
  OOWS Score on Day 28 | 0.6 (1.36) | 0.5 (0.87)
  Change from Baseline | -5.9 (3.19) | -5.9 (3.24)

6. Secondary Outcome: Addiction-related Severity Index (ASI-Lite): A Composite Score to Evaluate Seven Potential Problem Areas: Medical, Employment/Support Status, Alcohol, Drug, Legal, Family/Social, and Psychiatric
Description: The ASI-Lite is a standardized, multidimensional, semi-structured, comprehensive interview that estimates addiction-related problem severity profiles in seven domains commonly affected in substance abusers. ASI-lite composite score ranges from 0 (worst outcome) to 1 (best outcome) for each category. Reported here is the change in ASI-Lite from baseline to Day 28.
  The original drug use accounts for heroin, methadone, other opiates, analgesics, medicine/pills, cocaine, amphetamines, cannabis, hallucinogens, and inhalants. Modified drug use accounts for heroin, methadone, cocaine, and cannabis.
Time Frame: Baseline and 28 days
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Direct Suboxone Induction | Subutex-to-Suboxone Induction
Number analyzed (Participants) | 93 | 94
Score on a scale
  Medical | -0.05 (0.027) | -0.05 (0.027)
  Employment | -0.04 (0.034) | -0.02 (0.033)
  Employment satisfaction | -0.10 (0.030) | -0.01 (0.029)
  Alcohol use | -0.03 (0.017) | -0.01 (0.017)
  Drug use (Original) | -0.24 (0.018) | -0.23 (0.017)
  Drug use (Modified) | -0.36 (0.021) | -0.34 (0.021)
  Legal status | -0.09 (0.026) | -0.08 (0.025)
  Family/Social relations | -0.10 (0.040) | -0.10 (0.041)
  Other Family/Social relations | -0.08 (0.027) | -0.06 (0.026)
  Psychiatric | -0.12 (0.025) | -0.08 (0.024)

7. Secondary Outcome: Compliance Rate
Description: Compliance rate was calculated as the number of days study medication was taken divided by the number of days study medication should have been taken X 100. The number of days study medication should have been taken was equal to the duration of treatment.
Time Frame: 28 days
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Direct Suboxone Induction | Subutex-to-Suboxone Induction
Number analyzed (Participants) | 93 | 94
Percentage of days | 98.7 (4.22) | 98.4 (6.25)

8. Secondary Outcome: Responders at Day 28
Description: Responders were the number of participants in each group who received the scheduled 8- to 24-mg dose of Suboxone at study visit day. A participant who discontinued from the study was treated as a non-responder at the timepoint after the participant discontinued.
Time Frame: 28 days
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | Direct Suboxone Induction | Subutex-to-Suboxone Induction
Number analyzed (Participants) | 93 | 94
Participants
  Responder | 46 | 55
  Non-responder | 47 | 39

ADVERSE EVENTS:
Description: The population analyzed is the ITT population
Arm/Group | Direct Suboxone Induction | Subutex-to-Suboxone Induction
Serious Adverse Events (participants affected / at risk) | 1/93 | 3/94
Other Adverse Events (participants affected / at risk) | 61/93 | 64/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Direct Suboxone Induction (N=93) | Subutex-to-Suboxone Induction (N=94)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 1 (1)
EPILEPSY (Nervous system disorders) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
DRUG DEPENDENCE (Psychiatric disorders) | 1 (1) | 0 (0)
PERSONALITY DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Direct Suboxone Induction (N=93) | Subutex-to-Suboxone Induction (N=94)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 (5) | 4 (5)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 6 (7)
NAUSEA (Gastrointestinal disorders) | 8 (9) | 14 (15)
TOOTHACHE (Gastrointestinal disorders) | 6 (6) | 1 (1)
VOMITING (Gastrointestinal disorders) | 15 (16) | 11 (12)
ASTHENIA (General disorders) | 8 (8) | 5 (6)
CHILLS (General disorders) | 3 (3) | 6 (6)
FEELING COLD (General disorders) | 7 (7) | 10 (10)
MYALGIA (Musculoskeletal and connective tissue disorders) | 7 (8) | 11 (12)
HEADACHE (Nervous system disorders) | 7 (10) | 9 (10)
SOMNOLENCE (Nervous system disorders) | 10 (11) | 7 (9)
ANXIETY (Psychiatric disorders) | 19 (24) | 16 (17)
DRUG DEPENDENCE (Psychiatric disorders) | 16 (20) | 10 (15)
INSOMNIA (Psychiatric disorders) | 25 (27) | 26 (30)
RESTLESSNESS (Psychiatric disorders) | 8 (8) | 5 (6)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 22 (25) | 21 (25)
HOT FLUSH (Vascular disorders) | 5 (5) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI cannot publish an individual study until a publication disclosing results from multicenter studies is published. The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 45 days from the time submitted to the sponsor for review.